CLINICAL TRIAL: NCT00185211
Title: Open-label, Multi-center Phase III Extension of the Double-blind, Placebo-controlled BENEFIT Study (no. 92012/304747) to Obtain Long-term Follow-up Data of Patients With Clinically Definite Multiple Sclerosis (MS) and Patients With a First Demyelinating Event Suggestive of MS Treated With 8 MIU (250 µg) Interferon Beta-1b (Betaferon® / Betaseron®) Given Subcutaneously Every Other Day for at Least 36 Months.
Brief Title: BENEFIT Study (Betaferon® / Betaseron® in Newly Emerging Multiple Sclerosis for Initial Treatment) and BENEFIT Follow-up Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 91031; 305207 (Other: Company Internal)
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Results first posted 2010-11-30 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Initial IFNB-1b (Interferon beta-1b) (Experimental): Initial Betaferon/Betaseron treatment (Interferon beta-1b, IFNB-1b), 250 ug administered s.c. (subcutaneous) every other day, continued in Follow-up phase
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046)
- Initial Placebo (Experimental): Initial placebo treatment; Betaferon/Betaseron, 250 ug administered s.c. (subcutaneous) every other day offered in Follow-up phase (= this trial)
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046)

INTERVENTIONS:
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — Initial Betaferon/Betaseron treatment (Interferon beta-1b, IFNB-1b), 250 ug administered s.c. (subcutaneous) every other day, continued in Follow-up phase
  Arms: Initial IFNB-1b (Interferon beta-1b)
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — Initial placebo treatment; Betaferon/Betaseron, 250 ug administered s.c. (subcutaneous) every other day offered in Follow-up phase (= this trial)
  Arms: Initial Placebo

SUMMARY:
This study will primarily compare the long-term effects of an early and continued treatment with Betaferon/Betaseron (patients who were treated with active medication during the double-blind BENEFIT study) to treatment initiated either after Clinically Definite Multiple Sclerosis (CDMS) has been diagnosed or after two years (those patients who were treated with placebo during the double-blind BENEFIT study).

Analyses are based on the integrated data of the initial BENEFIT study and this follow-up study.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer HealthCare Pharmaceuticals Inc..

Bayer HealthCare Pharmaceuticals Inc. is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have reached scheduled end of study in BENEFIT, either by developing CDMS or by completing 24 months

Exclusion Criteria:

* No participation in the initial BENEFIT study

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 468 (Actual)
Dates: Start 2002-08; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (88):
- Austria (3):
  - Graz
  - Innsbruck
  - Vienna
- Belgium (4):
  - Brussels
  - Ghent
  - Leuven
  - Liège
- Canada (6):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Czechia (5):
  - Brno
  - Hradec Králové
  - Ostrava
  - Pilsen
  - Prague
- Glostrup Municipality, Denmark
- Finland (6):
  - Helsinki
  - Kuopio
  - Oulu
  - Seinäjoki
  - Tampere
  - Turku
- France (9):
  - Rennes, Brittany Region
  - Bordeaux, Gironde
  - Clermont-Ferrand
  - Dijon
  - Lille
  - Nancy
  - Nice
  - Paris
  - Toulouse
- Germany (20):
  - Ulm, Baden-Wurttemberg
  - München, Bavaria
  - Regensburg, Bavaria
  - Würzburg, Bavaria
  - Hennigsdorf, Brandenburg
  - Giessen, Hesse
  - Marburg, Hesse
  - Offenbach, Hesse
  - Braunschweig, Lower Saxony
  - Göttingen, Lower Saxony
  - Greifswald, Mecklenburg-Vorpommern
  - Cologne, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Homburg, Saarland
  - Halle, Saxony-Anhalt
  - Magdeburg, Saxony-Anhalt
  - Berlin, State of Berlin
  - Erfurt, Thuringia
- Hungary (3):
  - Szeged, Csongrád megye
  - Budapest
  - Debrecen
- Israel (2):
  - Haifa, Israel
  - Tel Litwinsky, Israel
- Italy (5):
  - Gallarate, Varese
  - Milan
  - Padua
  - Pavia
  - Torino
- Netherlands (2):
  - Sittard
  - Tilburg
- Bergen, Norway
- Poland (5):
  - Bydgoszcz
  - Krakow
  - Lodz
  - Lublin
  - Wroclaw
- Coimbra, Portugal
- Ljubljana, Slovenia
- Spain (7):
  - L'Hospitalet de Llobregat, Barcelona
  - Barakaldo, Vizcaya
  - Barcelona
  - Madrid
  - Málaga
  - Seville
  - Valencia
- Gothenburg, Sweden
- Switzerland (2):
  - Basel, Canton of Basel-City
  - Sankt Gallen
- United Kingdom (4):
  - Dundee, Scotland
  - Aberdeen
  - London
  - Sheffield

REFERENCES:
- [Background] Edan G, Kappos L, Montalban X, Polman CH, Freedman MS, Hartung HP, Miller D, Barkhof F, Herrmann J, Lanius V, Stemper B, Pohl C, Sandbrink R, Pleimes D; BENEFIT Study Group. Long-term impact of interferon beta-1b in patients with CIS: 8-year follow-up of BENEFIT. J Neurol Neurosurg Psychiatry. 2014 Nov;85(11):1183-9. doi: 10.1136/jnnp-2013-306222. Epub 2013 Nov 11. PMID 24218527
- [Background] Nagtegaal GJ, Pohl C, Wattjes MP, Hulst HE, Freedman MS, Hartung HP, Miller D, Montalban X, Kappos L, Edan G, Pleimes D, Beckman K, Stemper B, Polman CH, Sandbrink R, Barkhof F. Interferon beta-1b reduces black holes in a randomised trial of clinically isolated syndrome. Mult Scler. 2014 Feb;20(2):234-42. doi: 10.1177/1352458513494491. Epub 2013 Jul 10. PMID 23842212
- [Background] Penner IK, Stemper B, Calabrese P, Freedman MS, Polman CH, Edan G, Hartung HP, Miller DH, Montalban X, Barkhof F, Pleimes D, Lanius V, Pohl C, Kappos L, Sandbrink R. Effects of interferon beta-1b on cognitive performance in patients with a first event suggestive of multiple sclerosis. Mult Scler. 2012 Oct;18(10):1466-71. doi: 10.1177/1352458512442438. Epub 2012 Apr 4. PMID 22492127
- [Result] Kappos L, Freedman MS, Polman CH, Edan G, Hartung HP, Miller DH, Montalban X, Barkhof F, Radu EW, Metzig C, Bauer L, Lanius V, Sandbrink R, Pohl C; BENEFIT Study Group. Long-term effect of early treatment with interferon beta-1b after a first clinical event suggestive of multiple sclerosis: 5-year active treatment extension of the phase 3 BENEFIT trial. Lancet Neurol. 2009 Nov;8(11):987-97. doi: 10.1016/S1474-4422(09)70237-6. Epub 2009 Sep 10. PMID 19748319
- [Result] Hartung HP, Freedman MS, Polman CH, Edan G, Kappos L, Miller DH, Montalban X, Barkhof F, Petkau J, White R, Sahajpal V, Knappertz V, Beckmann K, Lanius V, Sandbrink R, Pohl C; BENEFIT Study Group. Interferon beta-1b-neutralizing antibodies 5 years after clinically isolated syndrome. Neurology. 2011 Aug 30;77(9):835-43. doi: 10.1212/WNL.0b013e31822c90d7. Epub 2011 Aug 17. PMID 21849647
- [Result] Freedman MS, Metzig C, Kappos L, Polman CH, Edan G, Hartung HP, Miller DH, Montalban X, Yarden J, Spector L, Fire E, Dotan N, Schwenke S, Lanius V, Sandbrink R, Pohl C. Predictive nature of IgM anti-alpha-glucose serum biomarker for relapse activity and EDSS progression in CIS patients: a BENEFIT study analysis. Mult Scler. 2012 Jul;18(7):966-73. doi: 10.1177/1352458511432327. Epub 2011 Dec 19. PMID 22183938
- [Result] Waschbisch A, Sandbrink R, Hartung HP, Kappos L, Schwab S, Pohl C, Wiendl H. Evaluation of soluble HLA-G as a biomarker for multiple sclerosis. Neurology. 2011 Aug 9;77(6):596-8. doi: 10.1212/WNL.0b013e318228c14d. Epub 2011 Jul 27. No abstract available. PMID 21795647
- [Result] Moraal B, Pohl C, Uitdehaag BM, Polman CH, Edan G, Freedman MS, Hartung HP, Kappos L, Miller DH, Montalban X, Lanius V, Sandbrink R, Barkhof F. Magnetic resonance imaging predictors of conversion to multiple sclerosis in the BENEFIT study. Arch Neurol. 2009 Nov;66(11):1345-52. doi: 10.1001/archneurol.2009.243. PMID 19901165
- [Result] Polman C, Kappos L, Freedman MS, Edan G, Hartung HP, Miller DH, Montalban X, Barkhof F, Selmaj K, Uitdehaag BM, Dahms S, Bauer L, Pohl C, Sandbrink R; BENEFIT investigators. Subgroups of the BENEFIT study: risk of developing MS and treatment effect of interferon beta-1b. J Neurol. 2008 Apr;255(4):480-7. doi: 10.1007/s00415-007-0733-2. Epub 2007 Nov 15. PMID 18004635
- [Result] Caloyeras JP, Zhang B, Wang C, Eriksson M, Fredrikson S, Beckmann K, Knappertz V, Pohl C, Hartung HP, Shah D, Miller JD, Sandbrink R, Lanius V, Gondek K, Russell MW. Cost-effectiveness analysis of interferon beta-1b for the treatment of patients with a first clinical event suggestive of multiple sclerosis. Clin Ther. 2012 May;34(5):1132-44. doi: 10.1016/j.clinthera.2012.03.004. Epub 2012 Apr 27. PMID 22541587
- [Result] Nielsen JM, Pohl C, Polman CH, Barkhof F, Freedman MS, Edan G, Miller DH, Bauer L, Sandbrink R, Kappos L, Uitdehaag BM. MRI characteristics are predictive for CDMS in monofocal, but not in multifocal patients with a clinically isolated syndrome. BMC Neurol. 2009 May 20;9:19. doi: 10.1186/1471-2377-9-19. PMID 19457248
- [Result] Barkhof F, Polman CH, Radue EW, Kappos L, Freedman MS, Edan G, Hartung HP, Miller DH, Montalban X, Poppe P, de Vos M, Lasri F, Bauer L, Dahms S, Wagner K, Pohl C, Sandbrink R. Magnetic resonance imaging effects of interferon beta-1b in the BENEFIT study: integrated 2-year results. Arch Neurol. 2007 Sep;64(9):1292-8. doi: 10.1001/archneur.64.9.1292. PMID 17846268
- [Result] Kappos L, Freedman MS, Polman CH, Edan G, Hartung HP, Miller DH, Montalban X, Barkhof F, Radu EW, Bauer L, Dahms S, Lanius V, Pohl C, Sandbrink R; BENEFIT Study Group. Effect of early versus delayed interferon beta-1b treatment on disability after a first clinical event suggestive of multiple sclerosis: a 3-year follow-up analysis of the BENEFIT study. Lancet. 2007 Aug 4;370(9585):389-97. doi: 10.1016/S0140-6736(07)61194-5. PMID 17679016
- [Result] De Jager PL, Chibnik LB, Cui J, Reischl J, Lehr S, Simon KC, Aubin C, Bauer D, Heubach JF, Sandbrink R, Tyblova M, Lelkova P; Steering committee of the BENEFIT study; Steering committee of the BEYOND study; Steering committee of the LTF study; Steering committee of the CCR1 study; Havrdova E, Pohl C, Horakova D, Ascherio A, Hafler DA, Karlson EW. Integration of genetic risk factors into a clinical algorithm for multiple sclerosis susceptibility: a weighted genetic risk score. Lancet Neurol. 2009 Dec;8(12):1111-9. doi: 10.1016/S1474-4422(09)70275-3. Epub 2009 Oct 29. PMID 19879194

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The full analysis set includes all 468 participants (particip.) with at least one administration of study drug in the placebo-controlled original study 92012, using treatment groups as randomized according to the minimization procedure regardless of the kind of study treatment (IFNB-1b/placebo) received. 19 subjects did not consent to the Follow-up
Period: Placebo-controlled Study (92012)
Arm/Group | Initial IFNB-1b (Interferon Beta-1b) | Initial Placebo
Started | 292 | 176
Completed | 271 | 166
Not Completed | 21 | 10
Not completed — Adverse Event | 8 | 0
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 9 | 7
Not completed — fulfilled local def. and McDonald crit. | 0 | 1
Not completed — Adverse event, then subject's withdrawal | 1 | 0
Period: Follow-up Study (91031 - This Study)
Arm/Group | Initial IFNB-1b (Interferon Beta-1b) | Initial Placebo
Started | 261 (10 of the 271 subjects completing the placebo-controlled study did not consent to the Follow-up.) | 157 (9 of the 166 subjects completing the placebo-controlled study did not consent to the Follow-up.)
Completed | 235 | 123
Not Completed | 26 | 34
Not completed — Adverse Event | 5 | 6
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 6 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 13 | 21
Not completed — other disease modif. treatment | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Initial IFNB-1b (Interferon Beta-1b) | Initial Placebo | Total
Number analyzed (Participants) | 292 | 176 | 468
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (7.6) | 30.7 (7.1) | 30.7 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 207 | 124 | 331
  Male | 85 | 52 | 137
Number of T2 lesions detected in screening MRI (Magnet-Resonance Imaging) [Number; unit: participants] — Only patients with at least two clinically silent lesions on the T2-weighted brain MRI scan with a size of at least 3 mm, at least one of which is ovoid or periventricular or infratentorial, were included. Number of T2 lesions with the three categories was used in the minimization procedure.
  participants
    2 to 4 T2 lesions | 42 | 25 | 67
    5 to 8 T2 lesions | 43 | 28 | 71
    at least 9 T2 lesions | 207 | 123 | 330
Number of participants with steroid use during the first clinical demyelinating event [Number; unit: participants] — The allocation of participants to the treatment arms was according to a minimization procedure with an element of randomization to minimize imbalances of treatment groups with respect to e.g. steroid use during first clinical demyelinating event. Steroid treatment was at the discretion of the investigator.
  participants
    Steroid Use | 209 | 123 | 332
    No Steroid Use | 83 | 53 | 136
Type of onset of disease (classification of first demyelinating event) [Number; unit: participants] — On the basis of the central classification of the patient's symptoms and signs, the first event was classified as either monofocal (a single central nervous system (CNS) lesion suffices to explain the patient's symptoms and signs) or multifocal (the patient's symptoms and signs can only be explained by multiple (i.e. more than one) CNS lesions.
  participants
    monofocal disease | 153 | 93 | 246
    multifocal disease | 139 | 83 | 222

OUTCOME MEASURES:

1. Primary Outcome: Time to Clinically Definite Multiple Sclerosis (CDMS) Represented by Kaplan-Meier Estimates of the Cumulative Percentage of Participants With CDMS at Selected Points in Time
Description: CDMS could be reached due to a qualifying relapse or sustained progression of 1.5 points on the expanded disability status scale (EDSS) as compared to the lowest EDSS obtained during screening or Day 1. The validity of CDMS diagnoses was confirmed by a central committee. The EDSS scale quantifies disability in MS in 8 functional systems, values vary between 0="normal neurological examination" and 10="death due to MS" measured in half-points on an ordinal scale. Time to CDMS = date of CDMS - date of Day 1 + 1 or time to CDMS = date of last clinical visit - date of Day 1 + 1 (right-censored)
Time Frame: up to 60 months after start of treatment
Population: The analysis followed the intention to treat (ITT) principle. After five years, in the initial placebo arm 94 participants and in the initial IFNB-1b arm 124 participants had reached CDMS diagnosis.
Measure: Number; unit: cum. percentage of particip. with CDMS
Arm/Group | Initial IFNB-1b (Interferon Beta-1b) | Initial Placebo
Number analyzed (Participants) | 292 | 176
cum. percentage of particip. with CDMS
  Kaplan-Meier estimate at year 2 | 26.9 | 45.0
  Kaplan-Meier estimate at year 3 | 36.7 | 51.2
  Kaplan-Meier estimate at year 5 | 46.2 | 57.3
Statistical Analysis 1: Comparison: Initial IFNB-1b (Interferon Beta-1b) vs Initial Placebo; The null hypothesis for comparison of initial IFNB-1b versus initial placebo treatment was: H0: The survival functions (i.e., the probability that time to CDMS is ≥ t) are identical for both treatment arms for all points in time t>0. The two-sided alternative hypothesis was: H1: The survival functions (i.e., the probability that time to CDMS is ≥ t) are not identical for both treatment arms for some points in time t>0; Test type: Superiority or Other; p = 0.0027, Log Rank — A 2-sided error level of 0.0253 was used for analyses at month 36 and 60 in order to keep the study-wise error level at 0.05. A conditional sequential testing approach was used for the family of null hypotheses of the primary efficacy variables
Statistical Analysis 2: Comparison: Initial IFNB-1b (Interferon Beta-1b) vs Initial Placebo; Time to CDMS was modelled by a Cox proportional hazards regression model with the following covariates: treatment group, steroid use during first event (yes vs. no), onset of disease (monofocal vs. multifocal) and number of T2 lesions at screening (categories: 2-4, 5-8 and at least 9 T2 lesions). The null hypothesis was: Initial IFNB-1b and initial placebo do not differ with regard to the hazard for CDMS, i.e. hazard ratio = 1; Test type: Superiority or Other; p = 0.0028, Regression, Cox; covariate adjustment: steroid use during first event, onset of disease, categorized number of T2 lesions at screening; Hazard Ratio (HR) = 0.663, 97.47% CI [0.488 to 0.902] — The direction of comparison is initial IFNB-1b (numerator) versus initial placebo (denominator), i.e. the Hazard Ratio represents the relative risk of initial IFNB-1b treatment compared to initial placebo treatment

2. Primary Outcome: Time to Confirmed Expanded Disability Status Scale (EDSS) Progression Represented by Kaplan-Meier Estimates of the Cumulative Percentage of Participants With Confirmed EDSS Progression at Selected Points in Time
Description: EDSS progression was defined as an increase in the expanded disability status scale (EDSS) of 1.0 point compared to the lowest EDSS score obtained during the screening or baseline visit, if this score was <= 5.5. A confirmed EDSS progression status was defined as an EDSS progression observed at two consecutive scheduled visits at least 140 days apart from each other. The EDSS scale is a method of quantifying disability in multiple sclerosis in eight functional systems and values vary between 0="normal neurological examination" and 10="death due to MS" measured in half-points on a scale.
Time Frame: up to 60 months after start of treatment
Population: The analysis followed the ITT principle. The 25%-percentile for time to confirmed EDSS progression was 908 days in the initial placebo arm but was not estimable in the initial IFNB-1b arm. After five years, in the initial placebo arm 47 participants and in the initial IFNB-1b arm 65 participants had reached confirmed EDSS progression.
Measure: Number; unit: percentage of particip. with EDSS progr.
Arm/Group | Initial IFNB-1b (Interferon Beta-1b) | Initial Placebo
Number analyzed (Participants) | 292 | 176
percentage of particip. with EDSS progr.
  Kaplan-Meier estimate at year 2 | 12.8 | 19.9
  Kaplan-Meier estimate at year 3 | 16.8 | 25.3
  Kaplan-Meier estimate at year 5 | 24.9 | 28.9
Statistical Analysis 1: Comparison: Initial IFNB-1b (Interferon Beta-1b) vs Initial Placebo; The null hypothesis for comparison of initial IFNB-1b versus initial placebo treatment was: H0: The survival functions (i.e., the probability that time to confirmed EDSS progression is ≥ t) are not identical for both treatment arms for some points in time t>0. The two-sided alternative hypothesis was: H1: The survival functions (i.e., the probability that time to confirmed EDSS progression is ≥ t) are identical for both treatment arms for some points in time t>0; Test type: Superiority or Other; p = 0.1768, Log Rank — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Initial IFNB-1b (Interferon Beta-1b) vs Initial Placebo; Time to confirmed EDSS progression was modelled by a Cox proportional hazards regression model with the following covariates: treatment group and volume of T2 lesions on screening MRI. The null hypothesis was: Initial IFNB-1b and initial placebo do not differ with regard to the hazard for confirmed EDSS progression, i.e. hazard ratio = 1; Test type: Superiority or Other; p = 0.1604, Regression, Cox; The variable used as additional covariate adjustment was volume of T2 lesions on screening MRI; Hazard Ratio (HR) = 0.764, 97.47% CI [0.497 to 1.174] — [estimate comment as in outcome 1, analysis 2]

3. Primary Outcome: Functional Assessment of Multiple Sclerosis (FAMS) Trial Outcome Index (TOI) at Month 60
Description: As an index of health related quality of life in people diagnosed with MS, the FAMS Trial Outcome Index covers overall physical health (sum of sub-scale scores Mobility, Symptoms, Thinking/Fatigue, Additional Concerns) with a score range from 0 to 148. A higher score reflects a higher overall physical health as reported by patients.
Time Frame: 60 months after start of treatment
Population: The analysis followed the ITT principle. Not all patients who completed the follow-up study could be included at month 60 as subject to copyright constraints and to the availability of validated language versions, FAMS assessments could not be conducted in all patients.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Initial IFNB-1b (Interferon Beta-1b) | Initial Placebo
Number analyzed (Participants) | 169 | 91
units on a scale | 125 [107 to 139] | 125 [104.83 to 140]
Statistical Analysis 1: Comparison: Initial IFNB-1b (Interferon Beta-1b) vs Initial Placebo; The null hypothesis H0: "The distribution of FAMS TOI at month 60, adjusted for baseline FAMS TOI, is identical for both treatment arms" was tested against the alternative hypothesis HA: "The distribution of FAMS TOI at month 60, adjusted for baseline FAMS TOI, is not the same in the two treatment arms" using a non-parametric analysis of covariance (ANCOVA); Test type: Superiority or Other; p = 0.8880, non-parametric ANCOVA — [p-value comment as in outcome 1, analysis 1]; Variable used as covariate: FAMS TOI measured at baseline
Statistical Analysis 2: Comparison: Initial IFNB-1b (Interferon Beta-1b) vs Initial Placebo; The null hypothesis H0: "The mean FAMS TOI at month 60, adjusted for baseline FAMS TOI, is identical for both treatment arms" was tested against the alternative hypothesis HA: "The mean FAMS TOI at month 60, adjusted for baseline FAMS TOI, is not the same in the two treatment arms" using a parametric analysis of covariance (ANCOVA); Test type: Superiority or Other; p = 0.3832, ANCOVA; Variable used as covariate: FAMS TOI measured at baseline

4. Secondary Outcome: Relapse-based Efficacy Domain: Time to Multiple Sclerosis (MS) According to McDonald Criteria
Description: MS according to the criteria by McDonald was reached if, in addition to the single clinical demyelinating event, both dissemination in space and dissemination in time were established by MRI-criteria or a new relapse. Time to McDonald MS is the difference of date of McDonald MS to the date of Day 1 + 1. For subjects without McDonald MS, time to McDonald MS is the difference from the maximum (date of last magnetic resonance imaging scan, date of last clinical visit) to the date of Day 1 + 1 (right-censored observation).
Time Frame: up to 60 months after start of treatment
Population: The analysis followed the ITT principle. After five years, in the initial placebo arm 151 participants and in the initial IFNB-1b arm 224 participants had reached McDonald MS diagnosis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Initial IFNB-1b (Interferon Beta-1b) | Initial Placebo
Number analyzed (Participants) | 292 | 176
months | 9.4 [8.8 to 12.1] | 6 [4.8 to 6.17]
Statistical Analysis 1: Comparison: Initial IFNB-1b (Interferon Beta-1b) vs Initial Placebo; The null hypothesis for comparison of initial IFNB-1b versus initial placebo treatment was: H0: The survival functions (i.e., the probability that time to McDonald MS is ≥ t) are identical for both treatment arms for all points in time t>0. The two-sided alternative hypothesis was: H1: The survival functions (i.e., the probability that time to McDonald MS is ≥ t) are not identical for both treatment arms for some points in time t>0; Test type: Superiority or Other; p = 0.000006, Log Rank — The two-sided error level for the exploratory analysis of the secondary outcome measures was of 0.05
Statistical Analysis 2: Comparison: Initial IFNB-1b (Interferon Beta-1b) vs Initial Placebo; Time to McDonald MS was modelled by a Cox proportional hazards regression model with the following covariates: treatment group, steroid use during first event (yes vs. no), onset of disease (monofocal vs. multifocal) and number of T2 lesions at screening (categories: 2-4, 5-8 and at least 9 T2 lesions). The null hypothesis was: Initial IFNB-1b and initial placebo do not differ with regard to the hazard for McDonald MS, i.e. hazard ratio = 1; Test type: Superiority or Other; p < 0.000001, Regression, Cox; covariate adjustment: steroid use during first event, onset of disease, categorized number of T2 lesions at screening; Hazard Ratio (HR) = 0.583, 95% CI [0.474 to 0.718] — The direction of comparison is initial IFNB-1b versus initial placebo, i.e. the Hazard Ratio represents the relative risk of initial IFNB-1b treatment compared to initial placebo treatment

5. Secondary Outcome: Relapse-based Efficacy Domain: Hazard Ratio for Recurrent Relapses
Description: A relapse was defined as the appearance of a new neurological abnormality or the reappearance of a neurological abnormality, separated by at least 30 days from onset of a preceding clinical demyelinating event. The time to the onset of recurrent relapses was determined for each subject according to the counting process representation for recurrent events. Time to a relapse was right-censored if a relapse-risk period ended without relapse. Based on the Andersen-Gill model the hazard ratio for recurrent relapses was estimated. Annualized relapse rates are provided as another outcome measure.
Time Frame: up to 60 months after start of treatment
Population: The analysis followed the Intention-To-Treat (ITT) principle. The hazard for recurrent relapses was modelled by an extension of the Cox Proportional Hazards (PH) regression model (Andersen-Gill Model).
Measure: Number; unit: Ratio
Groups:
- All Subjects: All subjects part of Intention-To-Treat (ITT) Population
Arm/Group | All Subjects
Number analyzed (Participants) | 468
Ratio | 0.797
Statistical Analysis 1: Comparison: All Subjects; The time to recurrent relapses was modelled by an extension of Cox's PH regression model (Andersen-Gill Model) for recurrent events with the following covariates: treatment group, steroid use during first event (yes vs. no), onset of disease (monofocal vs. multifocal) and number of T2 lesions at screening (2-4, 5-8 and at least 9 T2 lesions). The null hypothesis was: Initial IFNB-1b and initial placebo do not differ with regard to the hazard for recurrent relapses, i.e. hazard ratio = 1; Test type: Superiority or Other; p = 0.1265, Andersen-Gill Model — The two-sided error level for the exploratory analysis of the secondary outcome measures was of 0.05; Covariate adjustment: steroid use during first event, onset of disease, categorized number of T2 lesions at screening; Hazard Ratio (HR) = 0.797, 95% CI [0.595 to 1.066] — [estimate comment as in outcome 1, analysis 2]

6. Secondary Outcome: Relapse-based Efficacy Domain (Supportive): Annualized Relapse Rate
Description: The annualized relapse rate is defined as total number of relapses up to month 60 divided by the total observation time (last clinical visit minus first day of study treatment administration plus 1 of all participants) in years.
Time Frame: up to 60 months after start of treatment
Population: The analysis followed the ITT principle. For each treatment arm, the relapse rate is defined as total number of relapses up to month 60 divided by the total observation time in years.
Measure: Mean (95% Confidence Interval); unit: number of relapses per patient and year
Arm/Group | Initial IFNB-1b (Interferon Beta-1b) | Initial Placebo
Number analyzed (Participants) | 292 | 176
number of relapses per patient and year | 0.2139 [0.1895 to 0.2406] | 0.2695 [0.2337 to 0.3093]
Statistical Analysis 1: Comparison: Initial IFNB-1b (Interferon Beta-1b) vs Initial Placebo; Relapse rate was analyzed by a generalized linear Poisson regression model with individual relapse counts as dependent variable, covariates: treatment arm, steroid use during first event, onset of disease and categorized number of T2 lesions at screening and offset variable natural log of time (in years) as difference between last clinical visit and baseline visit. The treatment effect on the relapse rate was of primary interest; Test type: Superiority or Other; p = 0.0141, generalized linear Poisson regression — The two-sided error level for the exploratory analysis of the secondary outcome measures was of 0.05; covariate adjustment: steroid use during first event, onset of disease, categorized number of T2 lesions at screening; Risk Ratio (RR) = 0.7971, 95% CI [0.6650 to 0.9554] — The direction of comparison is initial IFNB-1b (numerator) versus initial placebo (denominator), i.e. the Risk Ratio represents the relative risk of initial IFNB-1b treatment compared to initial placebo treatment

7. Secondary Outcome: Disability-based Efficacy Domain: Multiple Sclerosis Functional Composite (MSFC) at Month 60
Description: The MSFC score consists of three sub-tests (Timed-25-Foot-Walk, 9-Hole-Peg-Test, 3" Paced Auditory Serial Addition Test [PASAT]). Standardized results (Z-scores) of the sub-tests and the overall MSFC Z-score as an average of the three Z-scores were derived using baseline data pooled over both treatment arms as reference population. Higher Z-scores reflect a better neurological status.
Time Frame: 60 months after start of treatment
Population: The analysis followed the ITT principle. Not all FAS patients completed the follow-up study or had MSFC results at month 60 available.
Measure: Median (Inter-Quartile Range); unit: Z-scores
Arm/Group | Initial IFNB-1b (Interferon Beta-1b) | Initial Placebo
Number analyzed (Participants) | 228 | 120
Z-scores | 0.226 [-0.163 to 0.502] | 0.225 [-0.207 to 0.619]
Statistical Analysis 1: Comparison: Initial IFNB-1b (Interferon Beta-1b) vs Initial Placebo; The null hypothesis H0: "The distribution of MSFC Z-scores at month 60 adjusted for baseline MSFC Z-score is identical for both treatment arms" was tested against the alternative hypothesis HA: "The distribution of MSFC Z-scores at month 60 adjusted for baseline MSFC Z-score is not the same in the two treatment groups" based on a non-parametric analysis of covariance (ANCOVA); Test type: Superiority or Other; p = 0.6078, non-parametric ANCOVA — The two-sided error level for the exploratory analysis of the secondary outcome measures was of 0.05; Variable used as covariate: MSFC Z-scores measured at baseline
Statistical Analysis 2: Comparison: Initial IFNB-1b (Interferon Beta-1b) vs Initial Placebo; The null hypothesis H0: "The mean MSFC Z-scores at month 60 adjusted for baseline MSFC Z-score are identical for both treatment arms" was tested against the alternative hypothesis HA: "The mean MSFC Z-scores at month 60 adjusted for baseline MSFC Z-score are not the same in the two treatment groups" based on a non-parametric analysis of covariance (ANCOVA); Test type: Superiority or Other; p = 0.8245, ANCOVA — The two-sided error level for the exploratory analysis of the secondary outcome measures was of 0.05; Variable used as covariate: MSFC Z-scores measured at baseline

8. Secondary Outcome: MRI (Magnet-Resonance Imaging)-Based Efficacy Domain: Cumulative Number of Newly Active Lesions at Month 60
Description: Newly active lesions are defined as displaying either new Gadolinium (Gd)-enhancement on T1-weighted scans or non-enhancement on T1-weighted scan but new on T2-weighted scan. The numbers of newly active lesions on yearly MRI scans were summed up to the cumulative number.
Time Frame: up to 60 months after start of treatment
Population: The analysis followed the ITT principle. Not all patients in the full analysis set completed the follow-up study or had MRI scan readings at month 60 available.
Measure: Median (Inter-Quartile Range); unit: cumulative number of lesions
Arm/Group | Initial IFNB-1b (Interferon Beta-1b) | Initial Placebo
Number analyzed (Participants) | 219 | 114
cumulative number of lesions | 4 [1 to 12] | 7 [2 to 18]
Statistical Analysis 1: Comparison: Initial IFNB-1b (Interferon Beta-1b) vs Initial Placebo; The null hypothesis H0: "The distribution of the cumulative number of newly active lesions at month 60 adjusted for the number of Gadolinium (Gd)-enhancing lesions on T1 at screening is identical for both treatment arms." was tested against the corresponding two-sided alternative hypothesis based on a non-parametric analysis of covariance (ANCOVA); Test type: Superiority or Other; p = 0.0062, non-parametric ANCOVA — The two-sided error level for the exploratory analysis of the secondary outcome measures was of 0.05; Variable used as covariate: number of Gd-enhancing lesions on T1 at screening
Statistical Analysis 2: Comparison: Initial IFNB-1b (Interferon Beta-1b) vs Initial Placebo; Assuming that the cumulative number of newly active lesions at month 60 follows a negative binomial distribution, a generalized linear model (logarithmic link function, covariate: number of Gd-enhancing lesions on T1 at BENEFIT screening) was set up in order to analyze the treatment effect on that MRI outcome; Test type: Superiority or Other; p = 0.0435, generalized linear model — The two-sided error level for the exploratory analysis of the secondary outcome measures was of 0.05; Distribution: negative binomial distribution; covariate: number of Gd-enhancing lesions on T1 at screening; Relative effect size = 0.7351, 95% CI [0.5436 to 0.9940] — The direction of comparison is initial IFNB-1b versus initial placebo

9. Secondary Outcome: MRI-based Efficacy Domain: Absolute Change of T2 Lesion Volume From Screening MRI to Month 60
Description: Absolute change of T2 lesion volume from screening MRI to month 60 was calculated as T2 lesion volume at month 60 minus T2 lesion volume at screening.
Time Frame: 60 months after start of treatment
Population: The analysis followed the ITT principle. Not all FAS patients completed the follow-up study or had MRI scan readings at month 60 available.
Measure: Median (Inter-Quartile Range); unit: cubic millimeter
Arm/Group | Initial IFNB-1b (Interferon Beta-1b) | Initial Placebo
Number analyzed (Participants) | 215 | 112
cubic millimeter | -123.0 [-849.0 to 240.0] | -194.5 [-657.5 to 367.5]
Statistical Analysis 1: Comparison: Initial IFNB-1b (Interferon Beta-1b) vs Initial Placebo; The null hypothesis H0: "The distribution of the absolute change of T2 lesion volume at month 60 adjusted for the T2 lesion volume at screening is identical for both treatment arms." was tested against the corresponding two-sided alternative hypothesis based on a non-parametric analysis of covariance (ANCOVA); Test type: Superiority or Other; p = 0.7801, non-parametric ANCOVA — The two-sided error level for the exploratory analysis of the secondary outcome measures was of 0.05; Variable used as covariate: T2 lesion volume at screening
Statistical Analysis 2: Comparison: Initial IFNB-1b (Interferon Beta-1b) vs Initial Placebo; The null hypothesis H0: "The mean absolute change of T2 lesion volume at month 60 adjusted for the T2 lesion volume at screening is identical for both treatment arms." was tested against the corresponding two-sided alternative hypothesis based on a parametric analysis of covariance (ANCOVA); Test type: Superiority or Other; p = 0.9408, ANCOVA — The two-sided error level for the exploratory analysis of the secondary outcome measures was of 0.05; Variable used as covariate: T2 lesion volume at screening

10. Secondary Outcome: MRI-based Efficacy Domain: Absolute Change of Volume of Black Holes From Screening MRI to Month 60
Description: Absolute change of volume of black holes from screening MRI to month 60 was calculated as volume of black holes at month 60 minus volume of black holes at screening.
Time Frame: 60 months after start of treatment
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: cubic millimeter
Arm/Group | Initial IFNB-1b (Interferon Beta-1b) | Initial Placebo
Number analyzed (Participants) | 217 | 114
cubic millimeter | 0 [-169 to 40] | 0 [-94 to 54]
Statistical Analysis 1: Comparison: Initial IFNB-1b (Interferon Beta-1b) vs Initial Placebo; The null hypothesis H0: "The distribution of the absolute change of volume of black holes at month 60 adjusted for the volume of black holes at screening is identical for both treatment arms." was tested against the corresponding two-sided alternative hypothesis based on a non-parametric analysis of covariance (ANCOVA); Test type: Superiority or Other; p = 0.6619, non-parametric ANCOVA — The two-sided error level for the exploratory analysis of the secondary outcome measures was of 0.05; Variable used as covariate: Volume of black holes at screening
Statistical Analysis 2: Comparison: Initial IFNB-1b (Interferon Beta-1b) vs Initial Placebo; The null hypothesis H0: "The mean absolute change of volume of black holes at month 60 adjusted for the volume of black holes at screening is identical for both treatment arms." was tested against the corresponding two-sided alternative hypothesis based on a parametric analysis of covariance (ANCOVA); Test type: Superiority or Other; p = 0.8558, ANCOVA — The two-sided error level for the exploratory analysis of the secondary outcome measures was of 0.05; Variable used as covariate: Volume of black holes at screening

11. Secondary Outcome: MRI-based Efficacy Domain: Percentage Change of Brain Volume From Screening MRI to Month 60
Description: Two-timepoint percentage brain volume change was estimated with Structural Image Evaluation, using Normalisation, of Atrophy (SIENA) software. The measurements describe the percentage change from screening in brain volume at month 60.
Time Frame: 60 months after start of treatment
Population: The analysis followed the ITT principle. Not all patients in the full analysis set completed the follow-up study or had MRI scan readings at month 60 available. There were several missing values in both treatment arms regarding the percentage brain volume change.
Measure: Median (Inter-Quartile Range); unit: Percentage of brain volume
Arm/Group | Initial IFNB-1b (Interferon Beta-1b) | Initial Placebo
Number analyzed (Participants) | 141 | 80
Percentage of brain volume | -2.281 [-3.672 to -1.062] | -1.771 [-3.294 to -0.667]
Statistical Analysis 1: Comparison: Initial IFNB-1b (Interferon Beta-1b) vs Initial Placebo; The null hypothesis H0: "The distribution of the percentage change of brain volume at month 60 adjusted for the brain volume at screening is identical for both treatment arms." was tested against the corresponding two-sided alternative hypothesis based on a non-parametric analysis of covariance (ANCOVA); Test type: Superiority or Other; p = 0.1208, non-parametric ANCOVA — The two-sided error level for the exploratory analysis of the secondary outcome measures was of 0.05; Variable used as covariate: Brain volume at screening
Statistical Analysis 2: Comparison: Initial IFNB-1b (Interferon Beta-1b) vs Initial Placebo; The null hypothesis H0: "The mean percentage change of brain volume at month 60 adjusted for the brain volume at screening is identical for both treatment arms." was tested against the corresponding two-sided alternative hypothesis based on a parametric analysis of covariance (ANCOVA); Test type: Superiority or Other; p = 0.0719, ANCOVA — The two-sided error level for the exploratory analysis of the secondary outcome measures was of 0.05; Variable used as covariate: Brain volume at screening

ADVERSE EVENTS:
Arm/Group | Initial IFNB-1b (Interferon Beta-1b) | Initial Placebo
Serious Adverse Events (participants affected / at risk) | 61/292 | 42/176
Other Adverse Events (participants affected / at risk) | 283/292 | 169/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial IFNB-1b (Interferon Beta-1b) (N=292) | Initial Placebo (N=176)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Accidental injury (Injury, poisoning and procedural complications) | 3 | 1
Allergic reaction (Immune system disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Cyst (General disorders) | 1 | 0
Fever (General disorders) | 0 | 1
Hernia (General disorders) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Mucous membrane disorder (General disorders) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Suicide attemp other than overdose (Psychiatric disorders) | 0 | 1
Surgery (Surgical and medical procedures) | 12 | 6
Unevaluable reaction (General disorders) | 10 | 8
Myocardial infarct (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Liver function test abnormal (Investigations) | 2 | 0
Goiter (Endocrine disorders) | 0 | 1
Thyroid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Injection site necrosis (General disorders) | 2 | 0
Injection site reaction (General disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Weight gain (Investigations) | 1 | 0
Bone fracture (not spontaneous) (Injury, poisoning and procedural complications) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 2 | 2
Emotional lability (Psychiatric disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Myoclonus (Nervous system disorders) | 1 | 0
Personality disorder (Psychiatric disorders) | 0 | 1
Psychosis (Psychiatric disorders) | 1 | 0
Psychotic depression (Psychiatric disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Multiple sclerosis (Nervous system disorders) | 11 | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 2
Breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Eye disorder (Eye disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 2
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Endometrial disorder (Reproductive system and breast disorders) | 0 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Initial IFNB-1b (Interferon Beta-1b) (N=292) | Initial Placebo (N=176)
Back pain (Musculoskeletal and connective tissue disorders) | 49 | 20
Asthenia (General disorders) | 89 | 53
Fever (General disorders) | 48 | 18
Flu syndrome (Infections and infestations) | 152 | 90
Pain (General disorders) | 36 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 33 | 15
Leukopenia (Blood and lymphatic system disorders) | 73 | 26
Injection site reaction (General disorders) | 163 | 71
SGOT increased (Investigations) | 34 | 7
SGPT increased (Investigations) | 50 | 14
Bilirubinemia (Hepatobiliary disorders) | 29 | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 29 | 20
Anxiety (Psychiatric disorders) | 33 | 18
Depression (Psychiatric disorders) | 56 | 41
Insomnia (Psychiatric disorders) | 37 | 21
Headache (Nervous system disorders) | 98 | 54
Multiple sclerosis (Nervous system disorders) | 112 | 82
Paresthesia (Nervous system disorders) | 82 | 53
Upper respiratory infection (Infections and infestations) | 96 | 59
Pharyngitis (Infections and infestations) | 47 | 26
Rash (Skin and subcutaneous tissue disorders) | 39 | 15
Abdominal pain (Gastrointestinal disorders) | 22 | 14
Accidental injury (Injury, poisoning and procedural complications) | 26 | 14
Allergic reaction (Immune system disorders) | 23 | 11
Chills (General disorders) | 17 | 5
Infection (Infections and infestations) | 29 | 11
Surgery (Surgical and medical procedures) | 22 | 14
Neck pain (Musculoskeletal and connective tissue disorders) | 11 | 9
Hypertension (Vascular disorders) | 13 | 9
Tooth disorder (Gastrointestinal disorders) | 19 | 9
Diarrhea (Gastrointestinal disorders) | 21 | 9
Gastroenteritis (Infections and infestations) | 19 | 14
Nausea (Gastrointestinal disorders) | 21 | 10
Vomiting (Gastrointestinal disorders) | 23 | 7
Liver function test abnormal (Investigations) | 19 | 6
Sore throat (Respiratory, thoracic and mediastinal disorders) | 19 | 11
Injection site pain (General disorders) | 24 | 9
Hyperglycemia (Metabolism and nutrition disorders) | 12 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 15
Muscle cramps (Musculoskeletal and connective tissue disorders) | 15 | 8
Myasthenia (Musculoskeletal and connective tissue disorders) | 16 | 10
Dizziness (Nervous system disorders) | 14 | 10
Hypertonia (Nervous system disorders) | 15 | 5
Vertigo (Ear and labyrinth disorders) | 10 | 10
Hypesthesia (Nervous system disorders) | 15 | 10
Bronchitis (Infections and infestations) | 27 | 15
Rhinitis (Infections and infestations) | 18 | 9
Sinusitis (Infections and infestations) | 19 | 16
Eye pain (Eye disorders) | 18 | 7
Abnormal vision (Eye disorders) | 17 | 8
Blurred vision (Eye disorders) | 17 | 4
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 15 | 12
Urinary tract infection (Infections and infestations) | 14 | 13

LIMITATIONS AND CAVEATS:
Participant Flow: Subject with "Other" as reason for not completing a study period are presented according to the NIH pre-specified categories as far as possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Submit for review any manuscript / abstract related to the Study at least 90 days prior to publication.The proposed publication / presentation shall only be made after BSP has obtained adequate patent protection for the Results, or after the patentable information has been taken out of the publication/presentation.